CLINICAL TRIAL: NCT01813786
Title: Clinical and Histological Evaluation of the 755nm Alexandrite Laser With Handpiece for the Treatment of Scars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cynosure, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Device Feasibility
Other Study IDs: CYN12-PICO-CAPHST-07
Record Dates: First submitted 2013-03-12; First posted 2013-03-19 (Estimated); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Scars
MeSH Terms: conditions — Cicatrix | interventions — Lasers, Solid-State

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 755nm Alexandrite Laser with Handpiece 2 (Experimental): Focusing energy on skin
  Interventions: Device: 755nm Alexandrite Laser with handpiece 2
- 755nm Alexandrite Laser with handpiece 3 (Experimental): Focusing energy on skin
  Interventions: Device: 755nm Alexandrite Laser with handpiece 3
- 755nm Alexandrite laser with handpiece 1 (Experimental): Focusing energy on skin
  Interventions: Device: 755nm Alexandrite Laser with handpiece 1

INTERVENTIONS:
Device: 755nm Alexandrite Laser with handpiece 2 — Focusing energy on skin
  Arms: 755nm Alexandrite Laser with Handpiece 2
Device: 755nm Alexandrite Laser with handpiece 1 — focusing energy at skin surface
  Arms: 755nm Alexandrite laser with handpiece 1
Device: 755nm Alexandrite Laser with handpiece 3 — Focusing energy on skin
  Arms: 755nm Alexandrite Laser with handpiece 3

SUMMARY:
Compare efficacy and safety of handpieces on the 755nm Alexandrite laser for the treatment of scars.

ELIGIBILITY:
Inclusion Criteria:

1. Is a healthy male or female between 18 and 85 years old
2. Has unwanted scars not including atrophic scars and wishes to undergo laser treatments.
3. Is willing to consent to participate in the study.
4. Is willing to comply with all requirements of the study including biopsies, being photographed, following post treatment care and attending all treatment and follow up visits.
5. Has Fitzpatrick skin types I to IV.

Exclusion Criteria:

1. The subject is female and pregnant, has been pregnant within the last 3 months, is currently breast feeding or planning a pregnancy during the study period.
2. The subject is hypersensitive to light exposure OR takes photo sensitized medication.
3. The subject has active or localized systemic infections.
4. The subject has a coagulation disorder or is currently using anti-coagulation medication (including but not limited to heavy aspirin therapy {greater than 81 mg per day}).
5. The subject has any condition which, in the investigator's opinion, would make it unsafe for the subject to participate in this research study.
6. The subject is currently enrolled in an investigational drug or device trial, or has received an investigational drug or been treated with an investigational device within 3 months prior to entering this study.
7. The subject has used Accutane within 6 months prior to enrollment.
8. The subject has the need to be exposed to artificial tanning devices or excessive sunlight during the trial.
9. The subject has had prior treatment with parenteral gold therapy (gold sodium thiomalate).
10. The subject has a history of keloids.
11. The subject has evidence of compromised wound healing.
12. The subject has a history of squamous cell carcinoma or melanoma.
13. The subject has a history of immunosuppression/immune deficiency disorders (including HIV infection or AIDS) or use of immunosuppressive medications.
14. The subjects has an allergy to lidocaine and epinephrine.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2012-12; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Subject Biopsy Sampling | 3 months post last treatment
  Histological examination of tissue samples will be compared between baseline and 3 months post treatment.

SECONDARY OUTCOMES:
Photographic evaluation as a measure of improvement. | up to 3 months post last treatment
  2D photographs to be taken at each visit and assessed at the end of the study by 2-3 blinded assessors for improvement.
Subject Biopsy Sampling | 2 weeks post treatment
  Histological examination of tissue samples will be compared between baseline and 2 weeks post treatment.
Subject Biopsy Sampling | 1 month post treatment
  Histological examination of tissue samples will be compared between baseline and 1 month post treatment.

OTHER OUTCOMES:
Number of participants with adverse events as a measure of safety and tolerability | up to 3 months post last treatment

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Krantz, Study Director — Cynosure, Inc.
Locations (1):
- Laser & Skin Surgery Center of New York, New York, New York, United States